CLINICAL TRIAL: NCT04964440
Title: Redo AF Sub Study (of the Pure EP 2.0 Main Study)
Status: Completed | Type: Observational
Sponsor: BioSig Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Redo AF Sub Study of Pure EP 2
Record Dates: First submitted 2021-07-02; First posted 2021-07-16 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation Recurrent
Keywords: reoccurring; repeat; revision; redo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- PURE EP Guided Procedures: Redo AF procedures guided by Pure EP System during an AF Ablation
  Interventions: Device: Pure-EP
- Standard Recording System Guided Procedures: Redo AF procedures guided by the Standard Recording System during an AF Ablation

INTERVENTIONS:
Device: Pure-EP — Advanced Signal Acquisition and Processing
  Groups: PURE EP Guided Procedures

SUMMARY:
This study is a sub study of the Pure EP 2.0 trial. In a redo atrial fibrillation population, this study is designed to collect pulmonary vein signals pre and post ablation therapy, along with other non-pulmonary vein signals of interest during a redo ablation procedure. These signals are later evaluated for clinical relevance and impact on the procedure.

DETAILED DESCRIPTION:
Cardiac electrophysiologists rely on the display of electrograms when performing EP studies and catheter ablations in patients with arrhythmias. To achieve effective outcomes without complications, it is vital that the recording system enables the recognition of clearly abnormal (scared myocardium) and normal electrical signals.

In a redo Atrial Fibrillation (AF) procedure, the patient had previously undergone an AF ablation procedure, but is still having AF episodes, which can be life threatening and have been shown to lead to strokes. Since the original AF procedure involved burning or freezing of myocardial tissue, this is now additional scar tissue and may cause more complex electrograms and intracardiac signals.

In this sub study, both the PURE EP™ system and the GE Cardiolab system will be running and recording signals during the entire procedure, with one of the systems displayed on the screen in the procedure room to guide the physician's decision-making. Even numbered subjects will be PURE EP™ guided and odd numbered subjected will be GE CardioLab guided. All other aspects of the procedure will proceed per standard of care. The study will be collect pulmonary vein signals pre and post ablation therapy, along with other non-pulmonary vein signals of interest during a redo ablation procedure.

After the physician has completed ablation treatment, matching signals of interest will be extracted from both the PURE EP™ system and the GE Cardiolab recording system as described in the main study. At a later date, a blinded electrophysiologist reviewer will evaluate the signals from both systems with a focus on tissue viability signals and the impact on the procedure. The survey results will then be compared to see the differences in clinical procedure decision-making based on the signal samples.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing scheduled elective cardiac ablation procedures who have signed an informed consent
2. Patients who are > 18 years of age.
3. Patients undergoing a repeat elective cardiac AF Procedure

Exclusion Criteria:

1. A complex arrhythmia secondary to a reversible cause
2. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
3. Any cardiac surgery within the past 60 days (2 months) (includes PCI)
4. Concurrent enrollment in a study evaluating another device or drug
5. A complex arrhythmia secondary to electrolyte imbalance, thyroid disease or non-cardiac issue
6. Presence of intra-cardiac thrombus or myxoma, interatrial baffle or patch, tumor or other abnormality that precludes catheter introduction or manipulation.
7. Presence of a condition that precludes vascular access.
8. Women of child baring potential whom are pregnant, lactating, or planning to become pregnant during the course of the clinical investigation.
9. Active illness or active systemic infection or sepsis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Atrial Fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
To assess the clinical procedure impact of PURE-EP signals of interest vs. a standard recording system in a Redo AF population | 6 months
  The signals of interest will undergo a homogenization process to remove all identifiers of the system used. At a later time, a blinded electrophysiologist reviewer will evaluate the signals for clinical relevance and procedural impact from both systems using the same Blinded Signal Assessment Form. The Blinded Assessment Form results will be compared to both each other and what was done at the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- St. David's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Collected intracardiac signal samples will be shared with the independent electrophysiologist reviewers, other physician investigators, and possibly other study collaborators like a biostatistician and clinical research organization
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The stored intracardiac signal samples from each enrolled subject will become available for review post-procedure and indefinitely.
Access Criteria: Access to the stored intracardiac electrogram signals will be determined and managed by BioSig Technologies.